CLINICAL TRIAL: NCT03284073
Title: First Clinical Live-Donor Uterus Transplantation Trial In Egypt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amro M. Hetta, M.Sc. (Other Government)
Collaborators: Al-Azhar University (Other); Mansoura University (Other)
Responsible Party: Sponsor-Investigator, Amro M. Hetta, M.Sc., Principal Investigator, Talkha Central Hospital
Organization: Talkha Central Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OG4
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Primary Uterine Infertility
Keywords: uterus; transplantation; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Human uterus transplantation from a live donor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterus Transplantation (Experimental): Patients undergo transplantation of the uterus from a live donor
  Interventions: Procedure: Uterus transplantation

INTERVENTIONS:
Procedure: Uterus transplantation — Transplantation of the uterus from a live donor and IVF treatment
  Other Names: UTx

SUMMARY:
More than a decade ago, uterus transplantation (UTx) as a highly experimental procedure was the treatment which had been developed for women suffering from absolute uterine factor infertility (AUFI) [uterus absence (congenital and surgical), or an abnormality (anatomic and functional)].

In Egypt, People's religions, current ethical and legal backgrounds make the option of live-donor uterus transplantation appealing rather than alternative pathways to parenthood. Thus, its clinical application for the first time in Egypt should be initiated after an extensive review and analysis of literature for UTx technology development in the world, and for further possible contributions to future prospects by Egypt proposed UTx project team which will participate in our study.

DETAILED DESCRIPTION:
More than a decade ago, uterus transplantation (UTx) as a highly experimental procedure was the treatment which had been developed for women suffering from absolute uterine factor infertility (AUFI) [uterus absence (congenital and surgical), or an abnormality (anatomic and functional)].

In Egypt, People's religions, current ethical and legal backgrounds make the option of live-donor uterus transplantation appealing rather than alternative pathways to parenthood. Thus, its clinical application for the first time in Egypt should be initiated after an extensive review and analysis of literature for UTx technology development in the world, and for further possible contributions to future prospects by Egypt proposed UTx project team which will participate in our study.

The study protocol includes live-donor UTx (mother, relative, friend) into women with AUFI. The recipient will be treated by standard immunosuppression and transfer of embryos (acquired by IVF before surgery) will be attempted after 8-12 months have passed from transplantation. Two official approvals must be obtained before starting recruitment process; from both (Higher Committee of Human Organ Transplantation of Egyptian Ministry of Health and Population, and Al-Azhar University Council).

ELIGIBILITY:
Inclusion Criteria:

* Less than 45 years old
* Good general health

Exclusion Criteria:

* Older than 45 years old
* Poor ovarian reserve
* Systematic or psychiatric disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 11 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Surviving transplants (8-12 months) | Up to 3 years after transplantation
  Follow up

SECONDARY OUTCOMES:
Spontaneous menstruation commencement | Up to 3 months after transplantation
  Observation
Pregnancy rate | Up to 3 years after transplantation
  IVF treatment
Live birth rate | Up to 4 years after transplantation
  IVF treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amro M. Hetta, M.Sc., Principal Investigator — Al-Azhar University
Locations (1):
- Mansoura Urology and Nephrology Center, Al Mansurah, Al-Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Scientific publications and Prospective thesis of MD Degree
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Background] Wei L, Xue T, Tao KS, Zhang G, Zhao GY, Yu SQ, Cheng L, Yang ZX, Zheng MJ, Li F, Wang Q, Han Y, Shi YQ, Dong HL, Lu ZH, Wang Y, Yang H, Ma XD, Liu SJ, Liu HX, Xiong LZ, Chen BL. Modified human uterus transplantation using ovarian veins for venous drainage: the first report of surgically successful robotic-assisted uterus procurement and follow-up for 12 months. Fertil Steril. 2017 Aug;108(2):346-356.e1. doi: 10.1016/j.fertnstert.2017.05.039. PMID 28778283
- [Background] Brannstrom M, Johannesson L, Bokstrom H, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Milenkovic M, Ekberg J, Diaz-Garcia C, Gabel M, Hanafy A, Hagberg H, Olausson M, Nilsson L. Livebirth after uterus transplantation. Lancet. 2015 Feb 14;385(9968):607-616. doi: 10.1016/S0140-6736(14)61728-1. Epub 2014 Oct 6. PMID 25301505
- [Background] Arnolds K, Gomez N, Berry A, Stadtlander K, Watson M, Tzakis A, Falcone T, Zimberg S. Assessment of an Alternative to the Uterine Vein for Venous Drainage in Human Uterine Transplantation: A Case Series Following Laparoscopic Hysterectomy. Gynecol Obstet Invest. 2016;81(5):436-41. doi: 10.1159/000442466. Epub 2016 Jan 22. PMID 26796796
- [Background] Molne J, Broecker V, Ekberg J, Nilsson O, Dahm-Kahler P, Brannstrom M. Monitoring of Human Uterus Transplantation With Cervical Biopsies: A Provisional Scoring System for Rejection. Am J Transplant. 2017 Jun;17(6):1628-1636. doi: 10.1111/ajt.14135. Epub 2017 Jan 3. PMID 27868389
- [Background] Fageeh W, Raffa H, Jabbad H, Marzouki A. Transplantation of the human uterus. Int J Gynaecol Obstet. 2002 Mar;76(3):245-51. doi: 10.1016/s0020-7292(01)00597-5. PMID 11880127
- [Background] Johannesson L, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Diaz-Garcia C, Olausson M, Brannstrom M. Uterus transplantation trial: 1-year outcome. Fertil Steril. 2015 Jan;103(1):199-204. doi: 10.1016/j.fertnstert.2014.09.024. Epub 2014 Oct 22. PMID 25439846
- [Background] Ghanem ME, El-Baghdadi LA, Badawy AM, Bakr MA, Sobhe MA, Ghoneim MA. Pregnancy outcome after renal allograft transplantation: 15 years experience. Eur J Obstet Gynecol Reprod Biol. 2005 Aug 1;121(2):178-81. doi: 10.1016/j.ejogrb.2004.11.035. PMID 16009483
- [Background] Jones BP, Saso S, Yazbek J, Smith JR. Uterine transplantation: past, present and future. BJOG. 2016 Aug;123(9):1434-8. doi: 10.1111/1471-0528.13963. Epub 2016 Mar 2. No abstract available. PMID 26931179
- [Background] Brannstrom M, Bokstrom H, Dahm-Kahler P, Diaz-Garcia C, Ekberg J, Enskog A, Hagberg H, Johannesson L, Kvarnstrom N, Molne J, Olausson M, Olofsson JI, Rodriguez-Wallberg K. One uterus bridging three generations: first live birth after mother-to-daughter uterus transplantation. Fertil Steril. 2016 Aug;106(2):261-6. doi: 10.1016/j.fertnstert.2016.04.001. Epub 2016 Apr 25. PMID 27125227
- [Background] Jarvholm S, Johannesson L, Clarke A, Brannstrom M. Uterus transplantation trial: Psychological evaluation of recipients and partners during the post-transplantation year. Fertil Steril. 2015 Oct;104(4):1010-1015. doi: 10.1016/j.fertnstert.2015.06.038. Epub 2015 Jul 28. PMID 26231464
- [Background] Jarvholm S, Johannesson L, Brannstrom M. Psychological aspects in pre-transplantation assessments of patients prior to entering the first uterus transplantation trial. Acta Obstet Gynecol Scand. 2015 Oct;94(10):1035-8. doi: 10.1111/aogs.12696. Epub 2015 Jun 30. PMID 26073658
- Available data/document: Study Protocol: NCT01844362 — http://clinicaltrials.gov